CLINICAL TRIAL: NCT04560647
Title: Pilot Studies Testing Levels of P63 in Psoriasis Skin Lesions
Status: Completed | Type: Observational
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Other Study IDs: 06956
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Psoriasis: Subjects diagnosed with psoriasis.
  Interventions: Other: No intervention - Psoriasis Subject
- Control: Subjects who do not have psoriasis.
  Interventions: Other: No intervention - Control Subject

INTERVENTIONS:
Other: No intervention - Psoriasis Subject — Not currently treated plaque psoriasis patients
  Groups: Psoriasis
Other: No intervention - Control Subject — Control subjects without plaque psoriasis and no family history of psoriasis
  Groups: Control

SUMMARY:
The purpose of this study is to understand the role of a specific protein, tumor protein p63 in the skin disease psoriasis. This study is to further understand how psoriasis lesions happens. An understanding of key mediators that lead to psoriasis might aid in the discovery of more effective treatments for this skin disorder. This is not an intervention study. The study is looking to obtain currently untreated plaque psoriasis biopsies and also biopsies from non psoriasis patients. Psoriasis and medical history will be collected then skin biopsies will be obtained from the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Female and Male adult subjects age 18 to 50 with plaque psoriasis that is currently untreated (no topical agents for 2 weeks, no systemic agents for 1 month) or controls w/o psoriasis and no family history of psoriasis.
* Must be able to give informed consent
* All skin types on Fitzpatrick Scale (Type I-VI)
* Able to provide medical history and list of medications for psoriasis and control subjects

Exclusion Criteria:

* Underlying diseases that could affect wound healing (e.g., uncontrolled diabetes mellitus)
* Tanning bed use within last 2 months
* Photodynamic Therapy or UVB treatments in past 2 months
* Female Subjects: pregnant or nursing
* History of abnormal scarring (i.e., keloids)
* Family history of psoriasis in first-degree relatives for control subjects

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Plaque psoriasis patients and control patients from the Dayton, OH area.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Abnormal P63 signaling levels | Day 0
  Determining if untreated psoriasis skin has abnormal p63 signaling

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Travers, MD, PhD, Principal Investigator — Wright State University
Locations (1):
- Wright State Physicians, Fairborn, Ohio, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT04560647/ICF_000.pdf